CLINICAL TRIAL: NCT03017586
Title: Subthalamic Nucleus (STN) and Globus Pallidus Internus (GPi) Deep Brain Stimulation (DBS) in Patients With Primary Dystonia（RELAX Study）
Brief Title: Efficacy and Safety of DBS in Patients With Primary Dystonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-023
Record Dates: First submitted 2017-01-05; First posted 2017-01-11 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STN (Experimental): DBS target with Subthalamic Nucleus (STN).
  Interventions: Device: Beijing Pins Medical Co., Ltd. Deep Brain Stimulator
- GPi (Experimental): DBS target with Globus Pallidus Internus (GPi).
  Interventions: Device: Beijing Pins Medical Co., Ltd. Deep Brain Stimulator

INTERVENTIONS:
Device: Beijing Pins Medical Co., Ltd. Deep Brain Stimulator — Deep Brain Stimulation for primary dystonia subjects

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of deep brain stimulation (DBS) of the subthalamic nucleus (STN) and globus pallidus internus (GPi) for primary dystonia.

DETAILED DESCRIPTION:
Dystonia is an uncommon brain disorder in which there is abnormal muscle tone producing twisting, writhing movements and abnormal postures. It is associated with abnormal electrical activity in two groups of nerve cells in the brain called the globus pallidus internus (GPi) and the subthalamic nucleus (STN). GPi DBS appears to be effective for medication-refractory focal and segmental dystonia affecting the cranial and cervical regions in open-label series, but recently GPi stimulation has been associated with subtle motor disturbances in previously non-dystonic body regions (i.e., arms and legs) in this population of patients. DBS of the STN has also been reported to be effective for treating generalized and cervical dystonia in small open label trials. STN DBS for cranial and cervical regions may provide similar efficacy in the treatment of dystonia as GPi DBS, but without unwanted stimulation-induced motor effects. Objectives of this study is to evaluate the safety and efficacy of STN-DBS and GPi-DBS for dystonia; Participants will be evaluated pre- and postoperatively with standard dystonia rating scales including the Burke-Fahn-Marsden Dystonia rating scale (BFMDRS), Changes in cognitive function will be assessed with neuropsychological testing. Stimulation parameters will be documented, and a patient questionnaire will be administered postoperatively to determine if patients are experiencing stimulation-induced motor adverse effects. Patient weight will be recorded at study visits. This pilot study will provide preliminary open label efficacy outcomes for STN DBS in the treatment of primary dystonia and will help determine if this target should be compared to GPi DBS in a larger double-blind trial.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory primary (systemic, segmental) dystonia diagnosed by a movement disorders neurologist
2. Severe functional impairment despite optimal medical management, including failed botulinum toxin therapy
3. Ability to follow up with post-operative study visits
4. Patients and their relatives have reasonable surgery expectations
5. Volunteer to participate in clinical trials, and signed consent form
6. Age 6-60 years

Exclusion Criteria:

1. Pregnancy or plan a pregnancy
2. Good treatment with Non-invasive therapy
3. Dopamine reactive dystonia ，Genetic degeneration ，Paroxysmal dystonia ，Secondary dystonia， Psychogenic dystonia
4. Brain MRI showing extensive brain atrophy or small vessel ischemic disease
5. Cognitive impairment(MMSE<24)
6. Severe depression or other serious mental illness
7. History of traumatic brain injury, tumor, or severe cerebrovascular disease
8. Severe brain atrophy (diagnosed by CT or MRI)
9. Hyperthermia therapy in implant parts
10. Abnormal in blood inspection, blood clotting disorders, liver and kidney dysfunction, or other clinical judgment cannot tolerate surgery
11. High blood pressure, serious heart diseases, or respiratory diseases
12. Diabetes
13. Long-term treatment of immunosuppressive or hormones
14. Implant pacemakers, defibrillators, cochlear and other nerve stimulators
15. Other diseases need frequent MRI examinations
16. Participated in any other clinical trials within 3 months
17. Reluctant or unable to implant surgery
18. Reluctant or unable to cooperate with follow-up
19. Other exclusion Criteria by researchers

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2020-09-13 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
change in Burke-Fahn-Marsden Dystonia Rating Scale (BFMDRS) movement score | 3，6 months

SECONDARY OUTCOMES:
Short-Form General Health Survey (SF-36) | 3，6 monthsthe Beck Anxiety Inventory31 (with scores ranging from 0 to 63 and higher scores indicating more severe anxiety)
  Quality of life was assessed with the Medical Outcomes Study 36-item Short-Form General Health Survey (SF-36), which evaluates both physical and mental components of functioning on a scale of 0 to 100, with higher scores indicating a higher level of function.
Visual analogue scale | 3，6 months
  The severity of dystonia and pain was assessed with the use of a visual analogue scale, with scores ranging from 0 to 10 and higher scores indicating greater severity
Measurements of walking | 3，6 months
  Measurements of walking (the duration and number of steps taken in a 14-m walk with one turn)
The Beck Depression Inventory | 3，6 months
  The Beck Depression Inventory (with scores ranging from 0 to 63 and higher scores indicating more severe depression)
Mini-Mental State Examination | 3，6 months
  Cognitive were assessed by mini-mental state examination
The rate of improvement of BFMDRS score | 3，6 months
  The rate of improvement of BFMDRS score that >25%、>50%、>75%

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Beijing Union Medical College Hospital, Beijing, Beijing Municipality
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Tongji Hospital of Tongji Univeristy, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital,School of Medicine,Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data is available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: De-identified data may be available after results have been published
Access Criteria: Individual participant data is available upon request.

REFERENCES:
- [Background] Benabid AL, Pollak P, Louveau A, Henry S, de Rougemont J. Combined (thalamotomy and stimulation) stereotactic surgery of the VIM thalamic nucleus for bilateral Parkinson disease. Appl Neurophysiol. 1987;50(1-6):344-6. doi: 10.1159/000100803. PMID 3329873
- [Background] Deep-Brain Stimulation for Parkinson's Disease Study Group; Obeso JA, Olanow CW, Rodriguez-Oroz MC, Krack P, Kumar R, Lang AE. Deep-brain stimulation of the subthalamic nucleus or the pars interna of the globus pallidus in Parkinson's disease. N Engl J Med. 2001 Sep 27;345(13):956-63. doi: 10.1056/NEJMoa000827. PMID 11575287
- [Background] Krack P, Pollak P, Limousin P, Hoffmann D, Xie J, Benazzouz A, Benabid AL. Subthalamic nucleus or internal pallidal stimulation in young onset Parkinson's disease. Brain. 1998 Mar;121 ( Pt 3):451-7. doi: 10.1093/brain/121.3.451. PMID 9549521
- [Background] Herzog J, Volkmann J, Krack P, Kopper F, Potter M, Lorenz D, Steinbach M, Klebe S, Hamel W, Schrader B, Weinert D, Muller D, Mehdorn HM, Deuschl G. Two-year follow-up of subthalamic deep brain stimulation in Parkinson's disease. Mov Disord. 2003 Nov;18(11):1332-7. doi: 10.1002/mds.10518. PMID 14639676
- [Background] Beric A, Kelly PJ, Rezai A, Sterio D, Mogilner A, Zonenshayn M, Kopell B. Complications of deep brain stimulation surgery. Stereotact Funct Neurosurg. 2001;77(1-4):73-8. doi: 10.1159/000064600. PMID 12378060
- [Background] Oh MY, Abosch A, Kim SH, Lang AE, Lozano AM. Long-term hardware-related complications of deep brain stimulation. Neurosurgery. 2002 Jun;50(6):1268-74; discussion 1274-6. doi: 10.1097/00006123-200206000-00017. PMID 12015845
- [Background] Umemura A, Jaggi JL, Hurtig HI, Siderowf AD, Colcher A, Stern MB, Baltuch GH. Deep brain stimulation for movement disorders: morbidity and mortality in 109 patients. J Neurosurg. 2003 Apr;98(4):779-84. doi: 10.3171/jns.2003.98.4.0779. PMID 12691402
- [Background] Benazzouz A, Piallat B, Pollak P, Benabid AL. Responses of substantia nigra pars reticulata and globus pallidus complex to high frequency stimulation of the subthalamic nucleus in rats: electrophysiological data. Neurosci Lett. 1995 Apr 14;189(2):77-80. doi: 10.1016/0304-3940(95)11455-6. PMID 7609923
- [Background] Benazzouz A, Gao DM, Ni ZG, Piallat B, Bouali-Benazzouz R, Benabid AL. Effect of high-frequency stimulation of the subthalamic nucleus on the neuronal activities of the substantia nigra pars reticulata and ventrolateral nucleus of the thalamus in the rat. Neuroscience. 2000;99(2):289-95. doi: 10.1016/s0306-4522(00)00199-8. PMID 10938434
- [Background] Dostrovsky JO, Levy R, Wu JP, Hutchison WD, Tasker RR, Lozano AM. Microstimulation-induced inhibition of neuronal firing in human globus pallidus. J Neurophysiol. 2000 Jul;84(1):570-4. doi: 10.1152/jn.2000.84.1.570. PMID 10899228
- [Background] Filali M, Hutchison WD, Palter VN, Lozano AM, Dostrovsky JO. Stimulation-induced inhibition of neuronal firing in human subthalamic nucleus. Exp Brain Res. 2004 Jun;156(3):274-81. doi: 10.1007/s00221-003-1784-y. Epub 2004 Jan 24. PMID 14745464
- [Background] Tai CH, Boraud T, Bezard E, Bioulac B, Gross C, Benazzouz A. Electrophysiological and metabolic evidence that high-frequency stimulation of the subthalamic nucleus bridles neuronal activity in the subthalamic nucleus and the substantia nigra reticulata. FASEB J. 2003 Oct;17(13):1820-30. doi: 10.1096/fj.03-0163com. PMID 14519661
- [Background] Hashimoto T, Elder CM, Okun MS, Patrick SK, Vitek JL. Stimulation of the subthalamic nucleus changes the firing pattern of pallidal neurons. J Neurosci. 2003 Mar 1;23(5):1916-23. doi: 10.1523/JNEUROSCI.23-05-01916.2003. PMID 12629196
- [Background] McIntyre CC, Grill WM, Sherman DL, Thakor NV. Cellular effects of deep brain stimulation: model-based analysis of activation and inhibition. J Neurophysiol. 2004 Apr;91(4):1457-69. doi: 10.1152/jn.00989.2003. Epub 2003 Dec 10. PMID 14668299
- [Background] Kupsch A, Benecke R, Muller J, Trottenberg T, Schneider GH, Poewe W, Eisner W, Wolters A, Muller JU, Deuschl G, Pinsker MO, Skogseid IM, Roeste GK, Vollmer-Haase J, Brentrup A, Krause M, Tronnier V, Schnitzler A, Voges J, Nikkhah G, Vesper J, Naumann M, Volkmann J; Deep-Brain Stimulation for Dystonia Study Group. Pallidal deep-brain stimulation in primary generalized or segmental dystonia. N Engl J Med. 2006 Nov 9;355(19):1978-90. doi: 10.1056/NEJMoa063618. PMID 17093249
- [Background] Vidailhet M, Vercueil L, Houeto JL, Krystkowiak P, Benabid AL, Cornu P, Lagrange C, Tezenas du Montcel S, Dormont D, Grand S, Blond S, Detante O, Pillon B, Ardouin C, Agid Y, Destee A, Pollak P; French Stimulation du Pallidum Interne dans la Dystonie (SPIDY) Study Group. Bilateral deep-brain stimulation of the globus pallidus in primary generalized dystonia. N Engl J Med. 2005 Feb 3;352(5):459-67. doi: 10.1056/NEJMoa042187. PMID 15689584
- [Background] Volkmann J, Wolters A, Kupsch A, Muller J, Kuhn AA, Schneider GH, Poewe W, Hering S, Eisner W, Muller JU, Deuschl G, Pinsker MO, Skogseid IM, Roeste GK, Krause M, Tronnier V, Schnitzler A, Voges J, Nikkhah G, Vesper J, Classen J, Naumann M, Benecke R; DBS study group for dystonia. Pallidal deep brain stimulation in patients with primary generalised or segmental dystonia: 5-year follow-up of a randomised trial. Lancet Neurol. 2012 Dec;11(12):1029-38. doi: 10.1016/S1474-4422(12)70257-0. Epub 2012 Nov 1. PMID 23123071
- [Background] Cao C, Pan Y, Li D, Zhan S, Zhang J, Sun B. Subthalamus deep brain stimulation for primary dystonia patients: a long-term follow-up study. Mov Disord. 2013 Nov;28(13):1877-82. doi: 10.1002/mds.25586. Epub 2013 Jul 16. PMID 23861342
- [Derived] Wang L, Shang H, Jin L, Xiong N, Hu X, Wang W, Liu Y, Yan J, Gao L, Wang Y, Wang Y, Fu P, Cai H, Zhang W, Xu S, Teng F, Ou R, Qiao L, Yang Y, Zhang M, Guo Y, Wan X. Subthalamic deep brain stimulation in isolated generalised or segmental dystonia (RELAX Study): a multicentre, randomised, double-blind, controlled trial. J Neurol Neurosurg Psychiatry. 2025 Oct 15;96(11):1077-1088. doi: 10.1136/jnnp-2025-335829. PMID 40480805

DOCUMENTS (1):
  • Study Protocol (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/86/NCT03017586/Prot_001.pdf